CLINICAL TRIAL: NCT03674255
Title: Use of Imaging and Blood Biomarkers to Improve the Diagnostic Accuracy of Cardiac Assessment by Stress Echocardiogram
Brief Title: Echocardiography: Value and Accuracy at REst and STress
Acronym: EVAREST
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Royal United Hospital Bath NHS Trust (Other); Tameside Hospital NHS Foundation Trust (Other); Royal Berkshire NHS Foundation Trust (Other Government); East Lancashire Hospitals NHS Trust (Other); Bradford Teaching Hospitals NHS Foundation Trust (Other Government); Calderdale and Huddersfield NHS Foundation Trust (Other); Great Western Hospitals NHS Foundation Trust (Other); Mid Essex Hospital NHS Trust (Other); Buckinghamshire Healthcare NHS Trust (Other); Wrightington, Wigan and Leigh NHS Foundation Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other); Milton Keynes University Hospital NHS Foundation Trust (Other Government); University Hospitals Bristol and Weston NHS Foundation Trust (Other); North Middlesex University Hospital (Other); Northumbria Healthcare NHS Foundation Trust (Other); London North West Healthcare NHS Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); Ultromics Ltd (Industry); National Institute for Health Research, United Kingdom (Other Government); King's College Hospital NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Poole Hospital NHS Foundation Trust (Other); Blackpool Teaching Hospitals NHS Foundation Trust (Other); Mid Yorkshire Teaching NHS Trust (Other); Northampton General Hospital NHS Trust (Other); North West Anglia NHS Foundation Trust (Unknown); Yeovil District Hospital NHS Foundation Trust (Other); East Suffolk and North Essex NHS Foundation Trust (Other); Nottingham University Hospitals NHS Trust (Other); Hampshire Hospitals NHS Foundation Trust (Other); Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: 18100
Record Dates: First submitted 2018-09-04; First posted 2018-09-17 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease; Ischaemic Heart Disease; Angina Pectoris
Keywords: Stress Echocardiography; Blood Biomarkers; Extracellular Vesicles; Imaging Biomarkers; Machine Learning; Artificial Intelligence; Ischaemic Heart Disease; Coronary Artery Disease; Angina Pectoris
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained from participants recruited into group 1. Samples will be obtained before and after the stress echocardiogram.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Participants in group 1 will be recruited at their stress echocardiogram appointment. Anonymised versions of the stress echocardiograms will be obtained, in addition to venous blood samples obtained from the cannula inserted as part of the standard clinical procedure. These blood samples will be collected before and after the stress echocardiogram. These participants will be followed up by telephone call after one year to determine whether they had any additional cardiac tests or events outside of their hospital trust. Medical records relating to the participant will be reviewed annually for up to 10 years to identify if the patient has been admitted and obtain health outcome data.
- 2: Participants in group 2 will be recruited at their stress echocardiogram appointment. Anonymised versions of the stress echocardiograms will be obtained. These participants will be followed up by telephone call after one year to determine whether they had any additional cardiac tests or events outside of their hospital trust. Medical records relating to the participant will be reviewed annually for up to 10 years to identify if the patient has been admitted and obtain health outcome data.
- 3: Participants in group 3 will be recruited at their stress echocardiogram appointment. Anonymised versions of the stress echocardiograms will be obtained. These participants will be followed up by telephone call after one year to determine whether they had any additional cardiac tests or events outside of their hospital trust. Medical records relating to the participant will be reviewed annually for up to 10 years to identify if the patient has been admitted and obtain health outcome data.
- 4: Participants in group 4 will be recruited at their stress echocardiogram appointment, regardless of the type of investigation. A simplified data set and an anonymised version of the stress echocardiography report will be collected as a part of this registry phase. Participants will be followed up over a 10-year period.

SUMMARY:
EVAREST will identify and validate novel blood and imaging biomarkers of potential value for consistent and accurate interpretation of stress echocardiography. During phase one, blood samples will be collected to assess the impact of cardiac stress on levels of circulating biomarkers and examine whether the measurement of these biomarkers can provide additional prognostic information. Phases one, two and three will also determine whether novel imaging biomarkers can be identified in the echocardiograms that can be used for objective interpretation of the stress echocardiograms. EVAREST will recruit up to 8000 patients (First 500 during phase one, an additional 500 during phase two and an additional 7000 during phase three) from multiple hospitals across United Kingdom, who have been referred for a stress echocardiogram as part of their investigations into ischaemic heart disease. Phase four of the study will continue into a clinical study cohort phase to capture information from all patients referred for a stress echocardiogram in the UK, regardless of the reason for investigation.This registry phase will run for 2 years, recruiting up to 15000 participants.

DETAILED DESCRIPTION:
Study Overview:

• Design

EVAREST is a multi-centre observational study comparing accuracy of novel quantitative stress echocardiography biomarkers for prediction of 12 month outcome against standard clinical interpretation.

• Scientific Justification

Coronary artery disease affects 2.3 million people in the UK and is responsible for 66 000 deaths each (BHF, 2018). As such, early diagnosis and intervention is crucial for saving lives and improving people's quality of life. Stress echocardiography is a commonly used, non-invasive imaging test used for detection of prognostically significant coronary artery disease. It allows the detection of regional wall motion abnormalities (RWMAs) which develop when the myocardium is not receiving adequate perfusion and, as such, indicates obstructive coronary artery disease. Average sensitivity and specificity for stress echocardiography is estimated at 81% and 82%, respectively (Geleijnse et al., 2009) in meta-analysis but remains highly subjective (Hoffmann et al., 1996) and subject to operator skill (Picano et al., 1991). Objective, quantifiable biomarkers in blood samples, or from images, acquired during the stress echocardiogram, which predict outcome of patients, could be used to reduce variability of stress echocardiography and ensure consistent and accurate results.

Aims

* To establish whether the measurement of specific blood biomarkers, in particular, extracellular vesicles, during a stress echocardiogram, can give additional prognostic information to stress echocardiography.
* To establish whether imaging biomarkers can provide additional prognostic information to stress echocardiography.

Phase One

Phase one will investigate the impact of cardiac stress on the levels of circulating biomarkers, in particular, extracellular vesicles. This phase will also assess whether they provide further prognostic information in addition to the echocardiogram. Blood samples will be collected from a cannula (inserted for the standard clinical procedure) before stress, during peak stress and during recovery and analysed to determine whether there were any changes in circulating extracellular vesicles during these three stages and whether these differ between patients with and without ischaemic heart disease.

Phase Two

Phase two continues recruitment for collection of stress echocardiogram images. Data collected during this phase will be compared with the data obtained during phase one to assess the usefulness of incorporating blood biomarkers into assessment of stress echocardiograms. In addition, the images obtained during phase two will be combined with the images collected during phase one to allow for the identification of novel imaging biomarkers which can be used to assist in the identification of patients with prognostically significant coronary disease.

Phase Three

Phase three will expand recruitment to allow evaluation of the generalisability of the imaging biomarkers identified in phase one and two across different healthcare settings, operators, stress protocols, machines and patient groups.

Phase Four

The fourth phase of the study allows for an assessment of all stress echocardiography practise in the UK and the demographics of patients being referred for stress echocardiogram. Phase four will investigate the use of stress echocardiography as a clinical procedure in the UK.

• Recruitment, Consent and Data Collection

Patients who have been scheduled a stress echocardiogram (using either pharmacological or exercise stress) as part of clinical investigations will be sent a participant information leaflet to read prior to their clinic appointment. When they are in the department, they will be approached by a study investigator to see whether they would be interested in taking part in the study and have the opportunity to ask the investigator any questions so that they fully understand the study. If they are interested in taking part, the process of obtaining informed consent will take place.

Following consent, the images acquired during the stress echocardiogram will be downloaded and anonymised with the participant's unique study ID number. These images will be transferred to the Oxford Research Echocardiography Core Laboratory (ORECL) for further analysis. Relevant medical history will be obtained for each participant as well as the clinician's interpretation of the echocardiogram. One year after the initial stress echocardiogram (range: 11-18 months), the participant will be followed-up to determine whether they underwent any further investigations for ischaemic heart disease (such as coronary angiography, cardiac magnetic resonance imaging, myocardial perfusion scintigraphy or repeat stress echocardiography) or had any coronary events. The participant may also be contacted via telephone to find out whether they were admitted to any other hospital for investigations. For phase one participants only, three blood samples (totalling approximately 40 ml) will be obtained before, at peak stress and after a recovery period, for the assessment of blood biomarkers. These samples will be taken through the cannula inserted as is routine during stress echocardiography. Participants will also give consent for follow-up information to be accessed for up to ten years after their initial stress echocardiogram.

• Outcome Assessment

Patient outcomes will be examined by an adjudication committee, blinded to the results of the stress echocardiograms. This committee will be led by a cardiologist and will examine all information obtained for a participant after the follow-up period has concluded. The criteria for confirming the presence of significant coronary artery disease include > 70% stenosis (assessed either via invasive coronary angiography or CT coronary angiography), an FFR < 0.85 or disease requiring intervention (either by percutaneous coronary intervention (PCI) or coronary artery bypass grafts (CABG)). Other end-points include coronary events (such as myocardial infarction) or death (attributed to coronary artery disease). If a patient has had no further investigations or events since their stress echocardiogram, their outcome will be recorded as normal.

• Confidentiality

All data obtained will be securely stored in accordance with the General Data Protection Regulations and Data Protection Act (2018) and Caldicott Principles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing a stress echocardiogram to investigate the presence of ischaemic heart disease (groups 1-3).
* Patients must be able to provide informed consent.
* Patients must be aged over 18 years of age.

Exclusion Criteria:

* Patients undergoing stress echocardiography to assess valvular function.
* Patients who are unwilling or unable to provide informed consent.
* Patients aged under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For phases 1 - 3, patients will be recruited when attending hospital for a stress echocardiogram to investigate the presence of ischaemic heart disease. For phase 4, patients attending hospital for a stress echocardiogram, for any investigation, will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 23000 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Prognostically Significant CAD | Data will be collected for ten years after the patient undergoes the stress echocardiogram.
  Patients will be followed up one year after their stress echocardiogram to determine whether they have prognostically significant CAD. This is defined as >70% stenosis assessed by angiography (either via invasive coronary angiography or CT coronary angiography), an FFR< 0.85 or the intention to revascularize (either via PCI or CABG). Any tests that occur in a ten year period after the stress echocardiogram will also be recorded.
Examination of Medical Records | Data will be collected for ten years after the patient undergoes the stress echocardiogram.
  Medical records will also be examined to check for any acute coronary syndromes within the year following the stress echocardiogram. Participants will also be contacted by telephone to capture any out-of-hospital events. Further follow-up data will be captured up to 10 years after the patient's initial stress echocardiogram.

SECONDARY OUTCOMES:
Quantification of Extracellular Vesicles (obtained from blood samples) by Flow Cytometry | Blood samples will be obtained before and after the stress echocardiogram. Analysis will be complete one year from the date of the stress echocardiogram
  The concentration of a comprehensive panel of cell-derived extracellular vesicles (such as erythrocyte, endothelial and platelet-derived extracellular vesicles) will be measured via flow cytometry in both the pre-stress and post-stress blood samples to assess the effect of cardiac stress on their concentration. The concentrations will also be compared between the patients with and without prognostically significant coronary artery disease to determine whether the concentration of extracellular vesicles is affected by coronary artery disease.
Assessment of Time to Diagnosis | Data will be collected for ten years after the patient undergoes the stress echocardiogram.
  We will assess whether the use of novel imaging and blood biomarkers can reduce the time to diagnosis of prognostically significant CAD.
Analysis of Potential Cost Savings Through the Use of Novel Biomarkers By the Reduction in Unnecessary Procedures | Data will be collected for ten years after the patient undergoes the stress echocardiogram.
  Health economic assessment will be carried out to determine whether the inclusion of imaging and blood biomarkers in the diagnostic process can ultimately lead to cost reductions through the reduction in unnecessary procedures and treatments.
Investigation into the use of stress echocardiography as a clinical procedure in the UK. | Data will be collected for ten years after the patient undergoes the stress echocardiogram.
  Analysis of the number and type of stress echocardiograms performed across UK NHS sites as well as demographic information on the patients referred for stress echocardiography and accuracy of stress echocardiography, using follow-up data.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Leeson, Principal Investigator — Cardiovascular Clinical Research Facility, University of Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsharqi M, Upton R, Mumith A, Leeson P. Artificial intelligence: a new clinical support tool for stress echocardiography. Expert Rev Med Devices. 2018 Aug;15(8):513-515. doi: 10.1080/17434440.2018.1497482. Epub 2018 Jul 19. No abstract available. PMID 29992841
- [Background] Augustine D, Ayers LV, Lima E, Newton L, Lewandowski AJ, Davis EF, Ferry B, Leeson P. Dynamic release and clearance of circulating microparticles during cardiac stress. Circ Res. 2014 Jan 3;114(1):109-13. doi: 10.1161/CIRCRESAHA.114.301904. Epub 2013 Oct 18. PMID 24141170
- [Background] Ayers L, Nieuwland R, Kohler M, Kraenkel N, Ferry B, Leeson P. Dynamic microvesicle release and clearance within the cardiovascular system: triggers and mechanisms. Clin Sci (Lond). 2015 Dec;129(11):915-31. doi: 10.1042/CS20140623. PMID 26359252